CLINICAL TRIAL: NCT00151866
Title: A Multicentre Randomised Study of the Efficacy of Transfusions With Platelets Stored in Platelet Additive Solution II Versus Plasma
Brief Title: Efficacy of Transfusions With Platelets Stored in Platelet Additive Solution II Versus Plasma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: P03.113
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2005-09

CONDITIONS: Hemato-Oncologic Patients; Myelosuppression; Thrombocytopenia
Keywords: Thrombopenia; Platelet transfusion; Increment; Transfusion reactions; Bleeding complication
MeSH Terms: conditions — Thrombocytopenia; Transfusion Reaction | interventions — Platelet Transfusion

INTERVENTIONS:
Procedure: platelet transfusion

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of transfusions with platelets stored in platelet additive solution II compared to plasma storage.

DETAILED DESCRIPTION:
Introduction: Utilization of platelet additive solutions (PASs) for storage of platelets has several advantages, however randomised studies testing the clinical efficacy are scarce. A prospective, randomised study comparing the efficacy of transfusions with platelets stored in Platelet Additive Solution II (PAS II) versus plasma showed that CCIs after transfusion with platelets stored in PAS II were significantly lower (1). Major drawbacks of this study were the exclusion of patients with clinical factors known to increase platelet consumption and a limited number of patients. A multicenter, randomised study to investigate clinical efficacy of platelets stored in PAS II versus plasma, also including patients with factors of increased platelet consumption, was performed. Methods: After consent patients > 18 years, without HLA- and/or HPA-alloantibodies, were randomised to receive pooled platelet concentrates (PC) suspended in either plasma or PAS II, leucoreduced, and stored up to 5 days. 1- and 24-hour CCI were the primary endpoints. Secondary endpoints were transfusion interval, adverse reactions and bleeding complications. An inclusion-period was defined as a maximum of 8 transfusions or 30 days after the first transfusion.

ELIGIBILITY:
Inclusion Criteria:patients > 18 years expected to receive platelet transfusions and informed consent -

Exclusion Criteria:HLA- and/or HPA- alloimmunization

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2003-10; Study Completion 2005-05

PRIMARY OUTCOMES:
Corrected count increment

SECONDARY OUTCOMES:
Bleeding complications

CONTACTS AND LOCATIONS:
Overall Officials: J.L.H. Kerkhoffs, MD, Principal Investigator — Sanquin rbbd
Locations (1):
- Leiden University Medical centre, Leiden, Netherlands